CLINICAL TRIAL: NCT06877195
Title: Multicenter Randomised Prospective Study for External Support Mesh VEST of Venous Coronary Grafts on the Right Territory: Mid-term Clinically Driven Re-rivascularization Events Comparison Between Sites Treated With VEST, Sites Treated With Bare Vein, Sites Treated With Other Conduits and de Novo Lesions on the Native Vessels
Brief Title: Multicenter Randomised Prospective Study for External Support Mesh VEST of Venous Coronary Grafts on the Right Territory
Acronym: RiVEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCRiVEST-1
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Cardiovascular Disease
Keywords: Coronary Artery Bypass Graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vested vein (Experimental): Usage of External mesh support (VEST) around the venous graft
  Interventions: Procedure: CABG
- Unvested vein (Active Comparator): Normally harvested and preserved "naked" vein used as a graft
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — Aortocoronary bypass procedures with venous grafts on right coronary territory

SUMMARY:
Multicentre randomised prospective study aimed at verifying medium-term patency of venous grafts on the right coronary artery territory, by clinical and/or instrumental follow-up with particular attention to clinically driven re-revascularisation events regarding the site of new lesions (granularly comparing sites already treated with VEST, sites treated with bare vein, sites treated with other conduits, de novo lesions on the native).

ELIGIBILITY:
Inclusion Criteria:

* combined or isolated interventions
* adequate vein calibre
* adequate graft flowmetry

Exclusion Criteria:

* inability to implant due to calibre disparity or inadequate flowmetry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Ri-revascularization of grafted territory | Till end of study (at least three years)
  Incidence of coronary ri-revascaularization by either angioplasty or surgical bypass concerning the grafted territory due to graft failure

SECONDARY OUTCOMES:
Major Cardiovascular and Cerebrovascular Events (MACCE) | Till end of study (at least three years)
  Incidence of Major Cardiovascular and Cerebrovascular Events

CONTACTS AND LOCATIONS:
Overall Officials: Luca Paolo Weltert, MD, Principal Investigator — Unicamillus
Locations (1):
- European Hospital, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonimized clinical parameters
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Form start to end of study
Access Criteria: Centers collaborating to active recruitment, to be added after the completion of their each institutional review